CLINICAL TRIAL: NCT04138849
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Safety, Pharmacokinetics and Pharmacodynamics of BBT-877 Following Single Doses in Healthy Japanese Male Subjects
Brief Title: Evaluate Safety, Pharmacokinetics and Pharmacodynamics of BBT-877 in Healthy Japanese Male
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bridge Biotherapeutics, Inc. (Industry)
Collaborators: KCRN Research, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BBT877-IPF-003
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Healthy Participants
MeSH Terms: interventions — ATX inhibitor BBT-877

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BBT-877 Low Dose (Experimental)
  Interventions: Drug: BBT-877 single dose
- BBT-877 Mid Dose (Experimental)
  Interventions: Drug: BBT-877 single dose
- BBT-877 High Dose (Experimental)
  Interventions: Drug: BBT-877 single dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo single dose

INTERVENTIONS:
Drug: BBT-877 single dose — Oral capsule, single dose.
  Arms: BBT-877 High Dose; BBT-877 Low Dose; BBT-877 Mid Dose
Drug: Placebo single dose — Oral capsule, single dose.
  Arms: Placebo

SUMMARY:
This study will collect safety, pharmacokinetic, and pharmacodynamic data in Japanese male subjects in order to support development worldwide.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent form as described in Appendix 3 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol
2. Healthy male 18 to 55 years of age inclusive at the time of signing the informed consent form
3. Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to dosing and throughout the study.
4. Overtly healthy as determined by medical evaluation including medical history, physical examination, clinical laboratory tests
5. Body mass index (BMI) within 18 to 30.0 kg/m2 (inclusive) and body weight not less than 50 kg
6. Blood pressure (after supine for 5 minutes) between 90 and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic.
7. A 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function.
8. Must agree to use contraception as detailed in Appendix 5 of this protocol during the treatment period and for at least 90 days after dosing of study treatment and refrain from donating sperm during this period
9. Be first generation Japanese.

Exclusion Criteria:

1. Has a history of or current clinically significant medical illness that the investigator considers should exclude the subject or that could interfere with the interpretation of the study results.
2. Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening and Day -1 as deemed appropriate by the investigator
3. Clinically significant abnormal physical examination, vital signs or 12 lead ECG at screening and Day -1 as deemed appropriate by the investigator
4. Has donated blood or had a significant blood loss (≤500 mL) within 8 weeks of Day 1 or history of anemia or history of decreased red blood cells (RBC).
5. Donated plasma within 7 days of Day -1
6. Estimated creatinine clearance <80 mL/min
7. Liver function tests (serum alkaline phosphatase [ALP], aspartate transaminase [AST], alanine aminotransferase [ALT]) and serum bilirubin (total and direct) 1.2 times above the upper limit of normal (ULN) at Screening or Day -1.
8. Baseline hemoglobin, hematocrit, red blood cell count below the lower limit of normal at Screening and Day -1.
9. Has a history of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV; has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at Screening.
10. History of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (4th edition) criteria within 5 years before screening or positive test result(s) for alcohol and/or drugs of abuse at screening and Day -1.
11. Positive cotinine test at Screening and Day -1.
12. History of presence of hypersensitivity or idiosyncratic reaction to the study drug(s) or related compounds.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | Up to Day 14.
  The number of AEs.

SECONDARY OUTCOMES:
Pharmacokinetics_AUC (the area under the curve) | Day 1 to Day 4
  AUC of BBT-877
Pharmacokinetics_Cmax (peak concentration) | Day 1 to Day 4
  Cmax of BBT-877
Pharmacodynamics_plasma LPA (Lysophosphatidic acid) | Day 1 to Day 4
  plasma LPA (18:2 and 20:4) concentrations over time and percent decrease from baseline LPA level

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Hyun Ryou, M.D., Ph.D., Study Director — Bridge Biotherapeutics, Inc.
Locations (1):
- WCCT, Cypress, California, United States